CLINICAL TRIAL: NCT04384484
Title: A Phase 3 Randomized Study of Loncastuximab Tesirine Combined With Rituximab Versus Immunochemotherapy in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma (DLBCL) (LOTIS-5)
Brief Title: Study to Evaluate Loncastuximab Tesirine With Rituximab Versus Immunochemotherapy in Participants With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Acronym: LOTIS 5
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADCT-402-311; 2020-000241-14 (EudraCT Number)
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Relapsed Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma
Keywords: Loncastuximab Tesirine; Refractory Diffuse Large B-Cell Lymphoma; Relapsed Diffuse Large B-Cell Lymphoma; Diffuse Large B-Cell Lymphoma; Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — loncastuximab tesirine; Rituximab; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Loncastuximab Tesirine + Rituximab (Lonca-R) (Experimental): Part 1 consists of a non-randomized safety run-in period evaluating the study drug for the first 20 participants.
  Participants will receive Lonca-R on Day 1 of each cycle for up to 8 cycles, where 1 cycle is 3 weeks. Lonca-R will be administered via an intravenous infusion of loncastuximab tesirine 150 µg/kg + rituximab 375 mg/m^2 Q3W for 2 cycles, then loncastuximab tesirine 75 µg/kg + rituximab 375 mg/m^2 Q3W for up to 6 additional cycles.
  Interventions: Drug: Loncastuximab Tesirine; Drug: Rituximab
- Part 2: Loncastuximab Tesirine + Rituximab (Lonca-R) (Experimental): Randomized participants will receive Lonca-R on Day 1 of each cycle for up to 8 cycles, where 1 cycle is 3 weeks. Lonca-R will be administered via an intravenous infusion of loncastuximab tesirine 150 µg/kg + rituximab 375 mg/m^2 every Q3W for 2 cycles, then loncastuximab tesirine 75 µg/kg + rituximab 375 mg/m^2 Q3W for up to 6 additional cycles.
  Interventions: Drug: Loncastuximab Tesirine; Drug: Rituximab
- Part 2: Standard Immunochemotherapy (R-GemOx) (Active Comparator): Randomized participants will receive R-GemOx consisting of rituximab, gemcitabine and oxaliplatin as a standard immunochemotherapy treatment on Day 1 or Day 2 of each cycle for up to 8 cycles, where 1 Cycle is 2 weeks. R-GemOx will be administered via an intravenous infusion of rituximab 375 mg/m^2 + gemcitabine 1000 mg/m^2 + oxaliplatin 100 mg/m^2 every 2 weeks (Q2W) for up to 8 cycles.
  Interventions: Drug: Rituximab; Drug: Gemcitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Loncastuximab Tesirine — Intravenous Infusion
  Other Names: Zynlonta; ADCT-402
  Arms: Part 1: Loncastuximab Tesirine + Rituximab (Lonca-R); Part 2: Loncastuximab Tesirine + Rituximab (Lonca-R)
Drug: Rituximab — Intravenous Infusion
Drug: Gemcitabine — Intravenous Infusion
  Arms: Part 2: Standard Immunochemotherapy (R-GemOx)
Drug: Oxaliplatin — Intravenous Infusion
  Arms: Part 2: Standard Immunochemotherapy (R-GemOx)

SUMMARY:
The purpose of this study is to evaluate the efficacy of loncastuximab tesirine (ADCT-402) combined with rituximab compared to standard immunochemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant aged 18 years or older
* Pathologic diagnosis of DLBCL, as defined by the 2016 World Health Organization classification (including participants with DLBCL transformed from indolent lymphoma), or high-grade B-cell lymphoma, with MYC and BCL2 and/or BCL6 rearrangements
* Relapsed (disease that has recurred following a response) or refractory (disease that failed to respond to prior therapy) disease following at least one multi-agent systemic treatment regimen [For China only: Adequate first line anti-DLBCL therapy is defined as having received at least 4 cycles of multiagent systemic treatment regimen containing rituximab and anthracycline, unless the participants are intolerant to the regimen, or had disease progression during the treatment. If disease progression occurred during the treatment period, then the disease is considered refractory where the number of treatment cycles will not be specified. For participants who are ineligible for anthracycline, anthracycline is not required.]
* Not considered by the investigator to be a candidate for stem cell transplantation based on performance status, advanced age, and/or significant medical comorbidities such as organ dysfunction
* Measurable disease as defined by the 2014 Lugano Classification as assessed by positron-emission tomography (PET)- computed tomography (CT) or by CT or magnetic resonance imaging (MRI) if tumor is not fluorodeoxyglucose (FDG)-avid on screening PET-CT
* Availability of formalin-fixed paraffin-embedded (FFPE) tumor tissue block (or minimum 10 freshly cut unstained slides if block is not available) Note: Any biopsy since initial diagnosis is acceptable, but if several samples are available, the most recent sample is preferred [For China only: This inclusion criterion is not applicable]
* ECOG performance status 0-2
* Adequate organ function as defined by screening laboratory values within the following parameters:

  1. Absolute neutrophil count ≥1000/μL (off growth factors for at least 72 hours)
  2. Platelet count ≥100000/μL without transfusion within the past 2 weeks
  3. ALT, AST, and GGT ≤2.5 × the upper limit of normal (ULN)
  4. Total bilirubin ≤1.5 × ULN (participants with known Gilbert's syndrome may have a total bilirubin up to ≤3 × ULN)
  5. Calculated creatinine clearance ≥30 mL/min by the Cockcroft and Gault equation

Note: A laboratory assessment may be repeated a maximum of two times during the Screening period to confirm eligibility.

* Negative beta-human chorionic gonadotropin (β-hCG) pregnancy test within 7 days prior to start of study drug (Cycle 1 Day 1) for women of childbearing potential
* Women of childbearing potential must agree to use a highly effective method of contraception from the time of giving informed consent until at least 12 months after the last dose of study treatment. Men with female partners who are of childbearing potential must agree to use a condom when sexually active or practice total abstinence from the time of giving informed consent until at least 7 months after the participant receives his last dose of study treatment.

Exclusion Criteria:

* Previous treatment with loncastuximab tesirine
* Previous treatment with R-GemOx
* Known history of hypersensitivity to a CD19 antibody, loncastumiximab tesirine (including SG3249) or any of its excipients, or history of positive serum human ADA to a CD19 antibody
* Pathologic diagnosis of Burkitt lymphoma
* Active second primary malignancy other than non-melanoma skin cancers, non-metastatic prostate cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast, or other malignancy that the Sponsor's medical monitor and Investigator agree and document should not be exclusionary
* Autologous transplant within 30 days prior to start of study drug (Cycle 1 Day 1)
* Allogeneic transplant within 60 days prior to start of study drug (Cycle 1 Day 1)
* Active graft-versus-host disease
* Post-transplantation lymphoproliferative disorders
* Active autoimmune disease, including motor neuropathy considered of autoimmune origin and other central nervous system (CNS) autoimmune disease
* Human immunodeficiency virus (HIV) seropositive with any of the following:

  1. CD4+ T-cell (CD4+) counts <350 cells/μL
  2. Acquired immunodeficiency syndrome-defining opportunistic infection within 12 months prior to screening
  3. Not on anti-retroviral therapy, or on anti-retroviral therapy for <4 weeks at the time of screening
  4. HIV viral load ≥400 copies/mL
* Serologic evidence of chronic hepatitis B virus (HBV) infection and unable or unwilling to receive standard prophylactic antiviral therapy or with detectable HBV viral load
* Serologic evidence of hepatitis C virus (HCV) infection without completion of curative treatment or with detectable HCV viral load
* History of Stevens-Johnson syndrome or toxic epidermal necrolysis
* Lymphoma with active CNS involvement, including leptomeningeal disease
* Clinically significant third space fluid accumulation (i.e., ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath)
* Breastfeeding or pregnant
* Uncontrolled hypertension (blood pressure ≥160/100 mm Hg repeatedly), unstable angina, congestive heart failure (greater than New York Heart Association class II), electrocardiographic evidence of acute ischemia, coronary angioplasty or myocardial infarction within 6 months prior to screening, uncontrolled atrial or ventricular cardiac arrhythmia, poorly controlled diabetes, severe chronic pulmonary disease, or other serious medical condition which is likely to significantly impair the participant's ability to tolerate the study treatment
* Major surgery within 4 weeks prior to start of study drug (Cycle 1 Day 1); radiotherapy, chemotherapy or other antineoplastic therapy within 14 days prior to start of study drug (Cycle 1 Day 1), except shorter if approved by the Sponsor
* Use of any other experimental medication within 14 days or 5 half-lives prior to start of study drug (Cycle 1 Day 1)
* Received live vaccine within 4 weeks of Cycle 1 Day 1
* Failure to recover to ≤Grade 1 (Common Terminology Criteria for Adverse Events [CTCAE] version 5.0) from acute non-hematologic toxicity (except alopecia) due to previous therapy prior to screening
* Congenital long QT syndrome or a corrected QTcF interval of ≥480 ms at screening (unless secondary to pacemaker or bundle branch block)
* Any other significant medical illness, abnormality, or condition that would, in the Investigator's judgment, make the participant inappropriate for study participation or put the participant at risk
* Known history of hypersensitivity to oxaliplatin or other platinum-based drugs, or gemcitabine, or rituximab, or any of their excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Up to 4 years

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 4 years
Overall Response Rate (ORR) | Up to 4 years
Complete Response Rate (CRR) | Up to 4 years
Duration of Response (DOR) | Up to 4 years
Number of Participants Who Experience At Least One Treatment-Emergent Adverse Event (TEAE) | Day 1 up to a maximum of Week 39
Number of Participants Who Experience At Least One Serious Adverse Event (SAE) | Up to 4 years
Number of Participants Who Experience a Clinically Significant Change From Baseline in Clinical Laboratory Results | Day 1 up to a maximum of Week 25
Number of Participants Who Experience a Clinically Significant Change From Baseline in Vital Sign Measurements | Day 1 up to a maximum of Week 25
Number of Participants Who Experience a Clinically Significant Change From Baseline in Physical Examinations | Day 1 up to a maximum of Week 25
Number of Participants Who Experience a Clinically Significant Change From Baseline in Eastern Cooperative Oncology Group (ECOG) Performance Status | Day 1 up to a maximum of Week 25
Number of Participants Who Experience a Clinically Significant Change From Baseline in Electrocardiogram (ECG) Results | Day 1 up to a maximum of Week 25
Average Concentration of Loncastuximab Tesirine at the End of Infusion | Day 1 of Cycles 1 through 6 (each cycle is 3 weeks)
Average Concentration of Loncastuximab Tesirine Before Infusion | Day 1 of Cycles 1 through 6 (each cycle is 3 weeks)
Number of Participants With Anti-Drug Antibody (ADA) Titers to Loncastuximab Tesirine | Day 1 up to a maximum of Week 25
Part 2: Change from Baseline in Health-Related Quality of Life (HRQoL) as Measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire -Core 30 (EORTC QLQ-C30) | Baseline up to a maximum of Week 25
Part 2: Change from Baseline in Health-Related Quality of Life (HRQoL) as Measured by the Lymphoma Subscale of Functional Assessment of Cancer Therapy- Lymphoma (LymS of FACT-Lym) | Baseline up to a maximum of Week 25
Part 2: Change from Baseline in Health-Related Quality of Life (HRQoL) as Measured by GP5 Item of the Functional Assessment of Cancer Therapy- Lymphoma (FACT-Lym) | Baseline up to a maximum of Week 25
Part 2: Change from Baseline in Health-Related Quality of Life (HRQoL) as Measured by EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) | Baseline to up to 4 years

CONTACTS AND LOCATIONS:
Locations (144):
- United States (11):
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Redlands Community Hospital, Redlands, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - UnityPoint Health - Iowa Oncology Research Association (IORA), Des Moines, Iowa
  - Norton Cancer Institute, Louisville, Kentucky
  - Comprehensive Cancer Centers of Nevada - Henderson, Las Vegas, Nevada
  - Kaiser Permanente Interstate Medical Office Central, Portland, Oregon
  - Hollings Cancer Center, Charleston, South Carolina
  - Virginia Cancer Specialists, Gainesville, Virginia
  - Medical College of Wisconsin Cancer Center Clinical Trials Office, Milwaukee, Wisconsin
- Argentina (4):
  - Clinica Adventista Belgrano, Belgrano, Buenos Aires
  - Clínica de Nefrología, Urología y Enfermedades Cardiovasculares S.A., Santa Fe, Buenos Aires
  - Instituto Médico Especializado Alexander Fleming, Buenos Aires, Distrito Federal
  - Grupo Gamma - Hospital Privado Rosario, Rosario, Santa Fe Province
- Belgium (4):
  - Algemeen Ziekenhuis Sint-Jan Brugge-Oostende - Campus Sint-Jan, Bruges
  - Cliniques Universitaires Saint-Luc, Brussels
  - Centre Hospitalier Universitaire Universite Catholique de Louvain, Namur
  - Algemeen Ziekenhuis Delta - Campus Rumbeke, Roeselare
- Brazil (10):
  - Hospital Erasto Gaertner - Liga Paranaense de Combate ao Câncer, Curitiba, Paraná
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Mãe de Deus - Centro Integrado de Oncologia, Porto Alegre, Rio Grande do Sul
  - Hospital do Câncer, Rio de Janeiro
  - Hemomed Instituto de Oncologia e Hematologia, São Paulo
  - A Beneficência Portuguesa de São Paulo - Unidade Mirante, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo
  - Hospital Santa Marcelina, São Paulo
- Canada (3):
  - Cross Cancer Institute, Edmonton
  - Research Institute of the McGill University Health Centre, Montreal
  - Hôpital Fleurimont, Sherbrooke
- Chile (3):
  - Centro de Estudios Clínicos SAGA, Santiago, Santiago Metropolitan
  - Instituto Oncológico Fundación Arturo López Pérez, Santiago, Santiago Metropolitan
  - CeCim - Centro de Estudios Clínicos e Investigaciones Médicas, Santiago, Santiago Metropolitan
- China (19):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Henan Cancer Hospital - Zhengzhou University, Zhengzhou, Henan
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China School of Medicine - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Chongqing University Cancer Hospital - Chongqing Cancer Hospital, Chongqing
  - Huizhou Municipal Central Hospital, Huizhou
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Institute of Hematology and Blood Diseases Hospital of CAMS - PUMC, Tianjin
  - Wuhan Union Hospital, Wuhan
  - Tongji Hospital, Wuhan
- Czechia (3):
  - Fakultni nemocnice Ostrava, Ostrava
  - Fakultni Nemocnice Kralovske Vinohrady, Prague
  - Fakultni nemocnice v Motole, Prague
- France (8):
  - Centre Hospitalier Regional Universitaire Brest, Brest, Brittany Region
  - Hôpital Avicenne, Bobigny
  - Centre Hospitalier Regional Universitaire Brest, Brest
  - Hôpital François Mitterrand, Dijon
  - Hôpital Privé du Confluent, Nantes
  - Hopital Universitaire Pitie Salpetriere, Paris
  - Hôpital Haut-Lévêque, Pessac
  - Centre de Lutte Contre le Cancer - Centre Henri-Becquerel, Rouen
- Hungary (4):
  - Heves Varmegyei Markhot Ferenc Oktatokorhaz es Rendelointezet, Heves, Budapest
  - Dél-pesti Centrumkórház - Országos Hematológiai és Infektológiai Intézet - Szent László, Budapest, Pest County
  - Semmelweis Egyetem, Budapest
  - Orszagos Onkologiai Intezet, Budapest
- Israel (7):
  - Samson Assuta Ashdod University Hospital, Ashdod
  - Soroka Medical Center, Beersheba
  - Shamir Medical Center (Assaf Harofeh), Be’er Ya‘aqov
  - Carmel Medical Center, Haifa
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva
  - The Chaim Sheba Medical Center, Tel Aviv
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (10):
  - Presidio Ospedaliero Universitario Santa Maria della Misericordia, Udine, Friuli Venezia Giulia
  - Azienda Socio Sanitaria Territoriale (ASST) degli Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliero - Universitaria Careggi, Florence
  - Ospedale Casa Sollievo della Sofferenza, Foggia
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST, Meldola
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Istituto Clinico Humanitas, Milan
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale San Raffaele, Milan
  - Istituto Europeo di Oncologia, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Sanitaria Locale della Romagna, Ravenna
- Japan (20):
  - National Hospital Organization - Nagoya Medical Center, Nagoya, Aichi-ken
  - Toyohashi Municipal Hospital, Toyohashi, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Matsuyama Red Cross Hospital, Matsuyama, Ehime
  - Gunma Prefectural Cancer Center, Ōta, Gunma
  - Sapporo Hokuyu Hospital, Sapporo, Hokkaido
  - Hokkaido Cancer Center, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Saitama Medical University - International Medical Center, Hidaka-Shi, Saitama
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Bunkyo-ku, Tokyo
  - National Hospital Organization Disaster Medical Center, Tachikawa, Tokyo
  - Fukushima Medical University Hospital, Fukushima
  - Gifu Municipal Hospital, Gifu
  - Kagoshima University Hospital, Kagoshima
  - Niigata University Medical and Dental Hospital, Niigata
  - National Hospital Organization Okayama Medical Center, Okayama
  - Osaka Prefectural Hospital Organization - Osaka International Cancer Institute, Osaka
- Mexico (6):
  - Boca Raton Clinical Research (BRCR) Global Mexico - Guadalajara, Guadalajara, Jalisco
  - PanAmerican Clinical Research Mexico - Guadalajara, Guadalajara, Jalisco
  - PanAmerican Clinical Research Mexico - Cuernavaca, Cuernavaca, Morelos
  - Hospital Universitario Dr. José Eleuterio González, Monterrey, Nuevo León
  - Hematológica Alta Especialidad, Huixquilucan
  - Boca Raton Clinical Research (BRCR) Global Mexico - Ciudad de México, Mexico City
- Netherlands (2):
  - Hagaziekenhuis Van Den Haag - Leyweg, The Hague, South Holland
  - Elisabeth-TweeSteden Ziekenhuis - Elisabeth, Tilburg
- Poland (8):
  - Pratia MCM Kraków, Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wrocławiu, Wroclaw, Lower Silesian Voivodeship
  - Szpitale Pomorskie Spółka Z Ograniczoną Odpowiedzialnością, Gdynia
  - Pratia Onkologia Katowice, Katowice
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz
  - Szpital Wojewódzki w Opolu, Opole
  - Centrum Medyczne Pratia Poznań, Skorzewo
  - Instytut Hematologii I Transfuzjologii, Warsaw
- Hospital Español Auxilio Mutuo, San Juan, Puerto Rico
- Spain (10):
  - Hospital del Mar - Parc de Salut Mar, Barcelona
  - Institut Català d'Oncologia - Hospital Duran i Reynals (ICO L'Hospitalet), Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Arnau de Vilanova, Valencia
- Istituto Oncologico della Svizzera Italiana, Bellinzona, Switzerland
- Turkey (Türkiye) (7):
  - Özel Koru Hastanesi, Çukurambar, Ankara
  - VKV Amerikan Hastanesi, Şişli, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi, Bornova, İzmir
  - Ondokuz Mayis Üniversitesi, Kurupelit, Samsun
  - Karadeniz Teknik Üniversitesi Tip Fakültesi, Ortahisar, Trabzon
  - Ankara Universitesi Tip Fakultesi - Cebeci Arastirma ve Uygulama Hastanesi, Ankara
  - Mehmet Kemal Dedeman Hematoloji Hastanesi, Kayseri
- United Kingdom (3):
  - The Royal Marsden NHS Foundation Trust, Sutton, England
  - NHS Greater Glasgow and Clyde, Glasgow
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No